CLINICAL TRIAL: NCT00408772
Title: Efficacy of Neoadjuvant XELOX/AVASTIN Therapy for Nonresectable Colorectal Liver Metastases With Secondary Hepatic Resection/Radiofrequency
Brief Title: Oxaliplatin, Capecitabine, and Bevacizumab Followed By Surgery and/or Radiofrequency Ablation in Patients With Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University of California, Davis (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200412546; UCDCC#131 (Other: University of California Davis); CDR0000517440 (Other: UC Davis)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin; Neoadjuvant Therapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Unresectable colorectal liver mets (Experimental)
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: oxaliplatin; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Procedure: radiofrequency ablation

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine
Drug: oxaliplatin
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. Giving chemotherapy and bevacizumab before surgery or radiofrequency ablation may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving oxaliplatin and capecitabine together with bevacizumab followed by surgery and/or radiofrequency ablation works in treating patients with colorectal cancer that has spread to the liver and cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the conversion rate of nonresectable disease to resectable disease in patients with nonresectable liver metastases secondary to colorectal adenocarcinoma treated with neoadjuvant therapy comprising oxaliplatin, capecitabine, and bevacizumab followed by hepatic resection and/or radiofrequency ablation.
* Evaluate progression-free survival of patients treated with this regimen.

Secondary

* Determine disease-free and overall survival of patients treated with this regimen.
* Determine the toxicities of this regimen in these patients.

OUTLINE:

* Neoadjuvant therapy: Patients receive oxaliplatin IV over 2 hours and bevacizumab IV over 1 hour on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for 4-6 courses in the absence of disease progression or unacceptable toxicity or until conversion to resectable disease.
* Surgery and/or radiofrequency ablation (RFA): Patients undergo hepatic resection (with or without RFA) when tumor is deemed resectable. Patients with stable (< 8 lesions) and unresectable disease undergo laparoscopic or percutaneous RFA. RFA repeats once 4-6 weeks later.
* Adjuvant therapy: Beginning 6-8 weeks after surgery and/or RFA, patients may receive adjuvant therapy comprising oxaliplatin, capecitabine, and bevacizumab, as in neoadjuvant therapy, for up to 4 courses.

After completion of study treatment, patients are followed every 4 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma metastatic to the liver

  * Unresectable liver metastases
* Measurable disease
* No evidence of extrahepatic metastases
* No CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 45 mL/min
* Urinary protein < 2+ by dipstick OR < 2 g by 24-hour urine collection
* Bilirubin < 2 times ULN
* SGOT and SGPT < 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 18 months after completion of study therapy
* Able to take oral medications (e.g., no dysphagia or malabsorption symptoms)
* No other prior malignancy unless in complete remission and off therapy for ≥ 5 years
* No known allergy to the study drugs
* No peripheral neuropathy > grade 1
* No uncontrolled infection
* No uncontrolled hypertension
* No active bleeding or hemoptysis
* No other serious concurrent illness within the past 12 months, including any of the following:

  * Nonstable coronary artery disease
  * Myocardial infarction
  * Transient ischemic attack
  * Cardiovascular accident

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* At least 28 days since prior major surgery
* Prior therapy for advanced disease allowed

  * No prior oxaliplatin-based therapy
* Concurrent maintenance and palliative treatment during study chemotherapy allowed (e.g., nutritional or transfusional support or pain control)
* No concurrent corticosteroids except when used under the following circumstances:

  * As oxaliplatin premedication
  * Anti-5-HT_3 as antiemetic
* No concurrent cold cap or iced mouth rinses
* No other concurrent chemotherapy
* No placement of hepatic artery port for regional chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Conversion rate of nonresectable disease to resectable disease | 48 months

SECONDARY OUTCOMES:
Disease-free and overall survival | 48 months
Objective response rate | 48 months
Duration of response | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Khatri, MD, FACS, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States